CLINICAL TRIAL: NCT07034131
Title: Improving Both Health in Women With the Use of Osteo-Buddy to Enhance Osteoporosis Knowledge - A Mixed Method Clinical Trial
Brief Title: Evaluation of Osteo-Buddy in Improving Osteoporosis Knowledge
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SingHealth Polyclinics (Other)
Responsible Party: Principal Investigator, Eunice Lim Shi Min, Family Physician, SingHealth Polyclinics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025-0064
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Osteoporosis Risk; Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): use of Osteo-Buddy for 4 weeks
  Interventions: Other: Osteo-Buddy; Other: Usual Care
- Control (Experimental): usual care - access to digitalised educational materials titled 'Healthy Bones'
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Osteo-Buddy — Osteo-Buddy is a Virtual Health Assistant (VHA) accessible on mobile phones that helps users with:
  1. Evaluating their risk level of osteoporosis
  2. Recommending screening and referrals
  3. Lifestyle interventions through motivation, education and tailored guidance
  As a 24/7 VHA, it offers real-time, personalised advice based on user inputs and health data.
  Arms: Intervention
Other: Usual Care — Access to digitalised educational materials on osteoporosis, titled 'Healthy Bones'

SUMMARY:
This is a pilot randomised controlled trial (RCT) to evaluate the use of a Virtual Health Assistant (VHA) named Osteo-Buddy in improving the knowledge of osteoporosis in older women.

DETAILED DESCRIPTION:
This study will involve evaluating the preliminary effectiveness and feasibility outcomes of the use of Osteo-Buddy, a Virtual Health Assistant (VHA), in improving the knowledge of osteoporosis in women aged 50 and above.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 and above
* Medium or high Osteoporosis Self-Assessment Tool for Asians (OSTA) score
* Not undertaken Bone Mineral Density (BMD) scan
* Never been treated with anti-osteoporosis medications such as bisphosphonates (e.g. alendronate, risendronate, ibandronate, zolendronate, pamidronate) or denosumab
* Able to read and speak English
* Currently use and own a smartphone where Osteo-Buddy can be used

Exclusion Criteria:

* Known terminal illness
* Visual, hearing and/or cognitive impairment or mental illness that renders them unable to provide informed consent

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Osteoporosis Prevention and Awareness Tool (OPAAT) score | On enrolment and 6-8 weeks post enrolment
  * 30-item questionnaire measuring osteoporosis knowledge
  * Minimum value = 0, maximum value = 30
  * Higher scores indicate a better outcome
System Usability Scale (SUS) | 6-8 weeks post enrolment
  * 10-item questionnaire assessing usability
  * Minimum value = 0, maximum value = 100
  * Higher scores mean a better outcome

SECONDARY OUTCOMES:
Recruitment rate | over the course of recruitment, estimated 3-4 months
  Percentage of participants successfully recruited among referred participants
Retention rate | 6-8 weeks post-enrolment
  Percentage of recruited participants who complete the study (return for 2nd visit and successfully complete 2nd questionnaire)
Utility rate | 4 weeks
  Percentage of intervention arm participants who utilise Osteo-Buddy over the 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eunice Lim, Principal Investigator — SingHealth Polyclinics

IPD SHARING:
Plan to Share IPD: No
In view of concerns regarding patient confidentaility and data security, IPD will not be shared.